CLINICAL TRIAL: NCT05981131
Title: QUILT-205: Long-Term Follow-Up of Subjects in QUILT-2.005 Phase 1b Trial of Intravesical N-803 Plus BCG in BCG-Naive Non-Muscle Invasive Bladder Cancer (NMIBC)
Brief Title: Follow up of Intravesical N-803 Plus BCG in BCG-Naive Non-Muscle Invasive Bladder Cancer (NMIBC)
Status: Active, not recruiting | Type: Observational
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: QUILT-205
Record Dates: First submitted 2023-07-18; First posted 2023-08-08 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Non Muscle Invasive Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — ALT-803; BCG Vaccine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: N803 plus Bacillus Calmette-Guerin (BCG) — QUILT-2.005 phase 1b (NCT02138734) was an open-label, dose-escalation, multicenter study of intravesical Bacillus Calmette-Guerin (BCG) plus N-803 in BCG-naïve non muscle invasive bladder cancer (NMIBC). A modified 3 + 3 design was used. Three subjects were enrolled at each dose level starting at 100 μg/instillation of N-803 and subsequently increasing to 200 μg/instillation and 400 μg/instillation. A standard dose of BCG, 50 mg, was employed. The primary endpoints of the study were: determination of the maximum tolerated dose (MTD) and designation of the recommended dose (RD) of N-803 in combination with BCG in subjects who have BCG-naïve NMIBC; safety profile of N-803 plus BCG in treated subjects; and disease response rate in treated subjects. A total of 9 subjects with high-risk, high-grade, BCG-naïve, NMIBC were enrolled into 3 cohorts and treated by intravesical administration of N-803 plus BCG.

SUMMARY:
The purpose of this clinical trial is to obtain long-term follow-up information and status of bladder cancer for patients who received study treatment in the QUILT-2.005 study.

DETAILED DESCRIPTION:
All 9 subjects that completed QUILT-2.005 phase 1b are planned to be enrolled in this study.

Thus, the maximum enrollment for this study is 9 subjects. All enrolled subjects will be followed every 12 months for life, or until withdrawal of consent, or if the Sponsor closes the study.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled and treated with intravesical N-803 plus BCG in the phase 1b portion of QUILT-2.005.

Exclusion Criteria:

* Not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who were enrolled and completed treatment with intravesical N-803 plus BCG in QUILT-2.005 phase 1b.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2023-08-17 (Actual); Primary Completion 2033-08-30 (Estimated); Study Completion 2033-08-30 (Estimated)

PRIMARY OUTCOMES:
Obtain Long Term Follow-Up data to be summarized using descriptive statistics | assessed up to 60 months
  Follow-up data on survival status, bladder cancer status (high-grade or low-grade), cystoscopy results (including number of cystoscopies done for each subject), biopsy results, upper tract evaluations, posttherapies and responses and outcomes of posttherapies, urine cytology results, and other medical history or treatments (if available) related to bladder cancer will be collected from subjects who were enrolled and treated in QUILT-2.005 phase 1b study with intravesical N-803 plus BCG.
  Study endpoints will be summarized with descriptive statistics. Continuous variables will be summarized as mean, median, standard deviation, and minimum and maximum values. Categorical variables will be summarized as the number and percentage of subjects in each category. All confidence intervals will be constructed at the two-sided 95% level of confidence.
Assess the Complete response yearly | assessed up to 60 months
  CR rate yearly following completion of QUILT-2.005 phase 1b for subjects with CIS disease with or without papillary disease at the initial diagnosis.
  CR rate (as determined by the Investigator) yearly following completion of QUILT-2.005 phase 1b will be reported along with a two-sided exact 95% confidence interval. The exact confidence interval will be calculated using the Clopper-Pearson method.
Asses Disease-free Survival | assessed up to 60 months
  To assess disease-free survival (DFS) since the first instillation of BCG plus N-803 in QUILT-2.005 phase 1b for subjects with papillary disease only at the initial diagnosis.
  DFS (as determined by the Investigator) will be analyzed using Kaplan-Meier (KM) analysis methods. Subjects that are disease-free at the end of follow-up with censored at the last disease-free assessment

CONTACTS AND LOCATIONS:
Overall Officials: Bobby Reddy, MD, Study Director — ImmunityBio, Inc.
Locations (1):
- Island Urology, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No